CLINICAL TRIAL: NCT01018797
Title: Intrastromal Corneal Ring Segment Implantation for High Astigmatism on Postkeratoplasty Eyes
Brief Title: Intrastromal Corneal Ring for High Astigmatism on Postkeratoplasty
Acronym: Anel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: BelquizRodrigues do Amaral Nassaralla, Instituto de Olhos de Goiânia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BQ-1-09-ARVO
Record Dates: First submitted 2009-11-21; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Astigmatism
Keywords: INTRASTROMAL CORNEAL RING; ASTIGMATISM; POSTKERATOPLASTY; EYES; To evaluate the clinical outcomes of ICRS implantation to correct high-degree astigmatism on eyes with prior penetrating keratoplasty (PK)
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- INTRASTROMAL CORNEAL RING SEGMENT (Experimental): Eighteen eyes of 18 patients, 8 men and 10 women, with high levels (> 5 diopters [D]) of postkeratoplasty astigmatism were studied in a nonrandomized, retrospective, observational case series. PK was performed to treat keratoconus in 15 patients, corneal scar after trauma in 2 patients, and Fuchs endothelial dystrophy in 1 patient.
  Interventions: Procedure: INTRASTROMAL CORNEAL RING SEGMENT

INTERVENTIONS:
Procedure: INTRASTROMAL CORNEAL RING SEGMENT — Corneal tunnels were created by means of mechanical dissection in all eyes. Intrastromal corneal ring segments implantation was indicated because of the existence of reduced best spectacle-corrected visual acuity (BSCVA) or contact lens intolerance.

SUMMARY:
To evaluate the clinical outcomes of Intrastromal Corneal Ring Segment (ICRS) implantation to correct high-degree astigmatism on eyes with prior penetrating keratoplasty (PK).

DETAILED DESCRIPTION:
Eighteen eyes of 18 patients, 8 men and 10 women, with high levels (> 5 diopters [D]) of postkeratoplasty astigmatism were studied in a nonrandomized, retrospective, observational case series. Mean age at the time of ICRS implantation was 38 years, range 22 to 49 years. PK was performed to treat keratoconus in 15 patients, corneal scar after trauma in 2 patients, and Fuchs endothelial dystrophy in 1 patient. All patients were spectacle and contact lens intolerant. There was no active corneal disease or problem apart from high astigmatism.

Minimum time of ICRS implantation was 2 years after PK and at least 6 months after sutures removal.

Preoperative examinations included personal medical ocular history, uncorrected visual acuity (UCVA), best spectacle-corrected visual acuity (BSCVA), refraction, keratometry, intraocular pressure (IOP) measurement by applanation tonometry, corneal astigmatism, surface regularity index, surface asymmetry index, tonometry, slit-lamp biomicroscopy, specular microscopy, and fundus examination.

Main outcome measures included UCVA, BSCVA, refraction, keratometry and computerized analysis of corneal topography.

All surgeries were performed by the same surgeon (BAN) at the Goiania Eye Institute, between July 2007 and January 2009. Corneal tunnels were created by means of mechanical dissection in all eyes. Intrastromal corneal ring segments implantation was indicated because of the existence of reduced best spectacle-corrected visual acuity (BSCVA) or contact lens intolerance. Intracorneal ring segments implantations were performed by the same surgeon following the same protocol. All eyes were implanted with the Cornealring (Visiontech Medical Optics, Belo Horizonte, MG, Brazil). Mean follow-up after ICRS implantation was 12 months (range, 09 to 22 months).

The procedure, its goals, and possible complications were explained and all patients signed an informed consent. The amount and axis of astigmatism to be corrected by ICRS was based on manifest refraction.

ELIGIBILITY:
Inclusion Criteria:

* > 5 diopters of postkeratoplasty astigmatism
* Patients 21 to 50 years old
* Conventional treatments have failed

Exclusion Criteria:

* Diabetes
* Autoimmune diseases

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, Study Chair — Instituto de Olhos de Goiânia
Locations (1):
- Instituto de Olhos de Goiânia, Goiânia, Goiás, Brazil